CLINICAL TRIAL: NCT06357195
Title: Implementation of DIAMOND-Lewy Guidelines for Emergency Department Antipsychotic Use in Older Patients With Cognitive and Movement Disorders
Brief Title: DIAMOND-Lewy Guidelines for Antipsychotic Use in Older Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Douglas Scharre, Professor of Clinical Neurology and Psychiatry, Division Director of Cognitive Neurology, Ohio State University
Other Study IDs: 2024H0075
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Emergency Psychiatric; Cognition Disorder; Movement Disorders; Antipsychotics and Neuroleptics Toxicity; Dementia With Lewy Bodies; Alteration in Mental Status; Behavior; Aging
MeSH Terms: conditions — Cognition Disorders; Movement Disorders; Lewy Body Disease; Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about current practices for the acute neuropsychiatric management of older adults during emergency department (ED) visits. Researchers will compare current standard of care practices with implemented guideline practice to see if standardized medication guidelines help reduce the usage of antipsychotics and/or benzodiazepines during acute presentations. The main questions this study aims to answer are:

* How many older adults are receiving antipsychotics or benzodiazepines during emergency department visits?
* Why are older adults receiving antipsychotics or benzodiazepines during emergency department visits?
* How many older adults who receive antipsychotics or benzodiazepines during emergency department visits have an underlying cognitive or movement disorder?
* What effects does administration of antipsychotics or benzodiazepines during emergency department visits have on patient outcomes in older adults and adults with neurocognitive disorders?
* Does implementation of standardized medication guidelines help reduce the usage of antipsychotics and/or benzodiazepines during acute presentations?

DETAILED DESCRIPTION:
Lewy Body Dementia (LBD) is the second most common type of dementia next to Alzheimer's Dementia, but many patients with this disease go undiagnosed or misdiagnosed. A clinical feature of this disease is sensitivity to certain medications such as antipsychotics and benzodiazepines, which can potentially worsen their symptoms and/or increase the risk of death. With neuropsychiatric symptoms being the leading cause for acute hospital visits in patients with LBD, over a third of patients receive antipsychotics in the hospital, a third end up needing a higher level of care after discharge, and a third of patients with dementia end up dying within the first year after an ED visit. Currently, there is not enough data for the best pharmacologic management of acute behavioral disturbances in older patients, but we do have international LBD guidelines that we can start to implement.

Since the ED is a place with high usage of antipsychotics/benzodiazepines, the purpose of this study is to measure the proportion of older patients who are receiving these medications during an ED visit. Of the older patients who received these medications, this study will measure which fraction of the patients might have an underlying diagnosis of dementia or movement disorder. The goal is to implement new hospital guidelines to help reduce the usage of these medications in older patients, thus the study will measure the proportion of older patients receiving these medications before and after the new hospital guidelines are implemented. The study will also directly measure the treatment knowledge of providers working in the ED by having them answer a clinical scenario/patient case question before and after the guidelines are presented to them. The ultimate goal of this study is to help improve patient outcomes in older people who visit the hospital by avoiding medications that could be potentially harmful to their health.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 54
* Received antipsychotic/benzodiazepine in the ED
* Have clinical signs or symptoms of underlying cognitive or movement disorders

Exclusion Criteria:

* None

Min Age: 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Older adults >54 years old who receive antipsychotics or benzodiazepines in the ED and older adults >54 years old who have underlying neurocognitive disorders and receive antipsychotics or benzodiazepines in the ED.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Antipsychotic/Benzodiazepine | From admission to discharge, up to 30 days
  Name of medication used
Clinical Indication | From admission to discharge, up to 30 days
  Reason for antipsychotic or benzodiazepine administration

SECONDARY OUTCOMES:
Length of Stay | From admission to discharge, up to 30 days
  Number of hours spent in the ED, number of days spent during hospital admission
Disposition | From admission to discharge, up to 30 days
  Discharge location order
Code Status | From admission to discharge, up to 30 days
  Resuscitation orders at the time of admission and discharge

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taylor JP, McKeith IG, Burn DJ, Boeve BF, Weintraub D, Bamford C, Allan LM, Thomas AJ, O'Brien JT. New evidence on the management of Lewy body dementia. Lancet Neurol. 2020 Feb;19(2):157-169. doi: 10.1016/S1474-4422(19)30153-X. Epub 2019 Sep 10. PMID 31519472
- [Background] Weintraub D, Chen P, Ignacio RV, Mamikonyan E, Kales HC. Patterns and trends in antipsychotic prescribing for Parkinson disease psychosis. Arch Neurol. 2011 Jul;68(7):899-904. doi: 10.1001/archneurol.2011.139. PMID 21747029
- [Background] Spears CC, Besharat A, Monari EH, Martinez-Ramirez D, Almeida L, Armstrong MJ. Causes and outcomes of hospitalization in Lewy body dementia: A retrospective cohort study. Parkinsonism Relat Disord. 2019 Jul;64:106-111. doi: 10.1016/j.parkreldis.2019.03.014. Epub 2019 Mar 23. PMID 30930058
- [Background] Hill JD, Schmucker AM, Siman N, Goldfeld KS, Cuthel AM, Chodosh J, Bouillon-Minois JB, Grudzen CR. Emergency and post-emergency care of older adults with Alzheimer's disease/Alzheimer's disease related dementias. J Am Geriatr Soc. 2022 Sep;70(9):2582-2591. doi: 10.1111/jgs.17833. Epub 2022 May 25. PMID 35612546
- [Background] Russek NS, Skappak C, Scheuermeyer F, Brousseau AA, McLeod SL, Melady D, Spencer M. Pharmacological Management of Agitation and Delirium in Older Adults: a Survey of Practices in Canadian Emergency Departments. Can Geriatr J. 2023 Sep 1;26(3):405-409. doi: 10.5770/cgj.26.666. eCollection 2023 Sep. PMID 37662063
- [Background] McKeith IG, Boeve BF, Dickson DW, Halliday G, Taylor JP, Weintraub D, Aarsland D, Galvin J, Attems J, Ballard CG, Bayston A, Beach TG, Blanc F, Bohnen N, Bonanni L, Bras J, Brundin P, Burn D, Chen-Plotkin A, Duda JE, El-Agnaf O, Feldman H, Ferman TJ, Ffytche D, Fujishiro H, Galasko D, Goldman JG, Gomperts SN, Graff-Radford NR, Honig LS, Iranzo A, Kantarci K, Kaufer D, Kukull W, Lee VMY, Leverenz JB, Lewis S, Lippa C, Lunde A, Masellis M, Masliah E, McLean P, Mollenhauer B, Montine TJ, Moreno E, Mori E, Murray M, O'Brien JT, Orimo S, Postuma RB, Ramaswamy S, Ross OA, Salmon DP, Singleton A, Taylor A, Thomas A, Tiraboschi P, Toledo JB, Trojanowski JQ, Tsuang D, Walker Z, Yamada M, Kosaka K. Diagnosis and management of dementia with Lewy bodies: Fourth consensus report of the DLB Consortium. Neurology. 2017 Jul 4;89(1):88-100. doi: 10.1212/WNL.0000000000004058. Epub 2017 Jun 7. PMID 28592453
- See also: DIAMOND-Lewy Management Toolkit — https://research.ncl.ac.uk/diamondlewy/managementtoolkit/